CLINICAL TRIAL: NCT05107635
Title: A Multicenter Patient Registry for Outcomes of Inappropriate Sinus Tachycardia and Postural Orthostatic Tachycardia Syndrome Treatment
Brief Title: Inappropriate Sinus Tachycardia Registry
Status: Recruiting | Type: Observational
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RP-2021-IST
Record Dates: First submitted 2021-10-28; First posted 2021-11-04 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Inappropriate Sinus Tachycardia; Postural Tachycardia Syndrome
Keywords: Inappropriate Sinus Tachycardia; Postural Tachycardia Syndrome;; Sinus Node Sparing Hybrid Procedure
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: AtriCure Commercially Available Devices — Epicardial and endocardial hybrid ablation procedure used to treat the IST or POTS using AtriCure commercially available devices.

SUMMARY:
The primary objective of this registry is to capture real-world safety and performance data on AtriCure devices used to ablate cardiac tissue when treating Inappropriate Sinus Tachycardia (IST) or Postural Tachycardia Syndrome (POTS). This is a retrospective and prospective, multicenter, US/OUS, observational data registry.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo or has undergone a procedure to treat IST or POTS using one or more AtriCure devices.
2. Subject is willing to provide written informed consent (defined as legally effective, documented confirmation of a subject's voluntary agreement to participate in this Registry) or authorization per institution and geographical requirements

Exclusion Criteria:

1. Subject is enrolled in a concurrent study that may impact treatment outcome of IST or POTS.
2. Subject with exclusion criteria required by FDA or local governance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The IST registry eligibility is open to sites and physicians performing the described treatments for patients diagnosed with IST and POTS. Subjects must have been scheduled to undergo or have undergone the described treatments for IST or POTS by their physicians. Registry participating sites will enroll patients that meet all inclusion criteria and no exclusion criteria without preselection or bias.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
AtriCure commercially available devices used to treat IST or POTS | 12 months
  The IST Registry will attempt to enroll all eligible patients at registry sites who have already had or are scheduled to have a procedure to treat IST/POTS that includes the use of at least one commercially available AtriCure cardiac ablation devices.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Stanford University, Palo Alto, California
  - Sequoia Hospital, Redwood City, California
  - University of Florida, Gainesville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Kansas City Cardiac Arrhythmia Research, Kansas City, Kansas
  - MedStar Health Research Institute, Hyattsville, Maryland
  - The Carl & Edyth Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Intermountain Medical Center, Murray, Utah
- Universitair Ziekenhuis Brussels, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No